CLINICAL TRIAL: NCT00192192
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Investigate Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold Adapted (CAIV-T) in Healthy Adults Aged 18 to 64 Years
Brief Title: Trial to Investigate Immune Responses Elicited by a Liquid Formulation of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold Adapted (CAIV-T) in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D153 P001
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2006-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

INTERVENTIONS:
Biological: CAIV-T

SUMMARY:
To perform a variety of assays on blood, serum, nasal wash samples and cells obtained from healthy adult subjects for the purposes of developing assays for application in the further investigation of immune responses generated by influenza virus vaccine, trivalent, types A and B, live, cold-adapted (liquid CAIV-T; Wyeth Lederle Vaccines, Marietta, PA).

ELIGIBILITY:
Inclusion Criteria:

* who are between 18 to 64 years of age. Subject must be at least 18 years of age and no older than 64 years of age at the time informed consent is obtained;
* eligible female subjects, who are of childbearing potential, who have a negative urine pregnancy test results prior to study vaccination. Females who are surgically sterile or post-menopausal do not require pregnancy testing.
* who are determined by medical history, physical examination and clinical judgement to be eligible for this study. Subjects with stable pre-existing disease, defined as disease not requiring change in therapy or hospitalization within 12 weeks before receipt of study vaccination will be eligible.
* who have provided written informed consent after the nature of the study has been explained;
* who, will be available for two month duration of the trial (from enrollment to study completion);
* who can be reached by study staff for the post-vaccination contact [telephone, clinic or home visit]

Exclusion Criteria:

* who are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; or cytotoxic agents;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* have an immunosuppressed or an immunocompromised individual living in the same household;
* with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine or placebo;
* who were administered any live virus vaccine within one month prior to enrollment;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* who, received a dose of influenza treatment (commercial or investigational) one month prior to enrollment. The prophylactic use of influenza antivirals is not permitted.
* who receive any influenza vaccine in the 6 months prior to enrollment, or a non-study influenza vaccine since enrollment;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results; Note: A pregnant household member is not considered a contraindication to enrollment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2000-11; Study Completion 2000-12

PRIMARY OUTCOMES:
Assays on blood, serum, nasal wash samples and cells obtained from healthy adult subjects

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (1):
- Stamford Hospital, Stamford, Connecticut, United States